CLINICAL TRIAL: NCT00813761
Title: Clinical Evaluation of the Long-Term Effects of Contact Lens Care Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-4522
Record Dates: First submitted 2008-12-17; First posted 2008-12-23 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 02Optix CL and ReNu MPS with SICS (Other): O2Optix contact lens and ReNu MultiPlus Multi-Purpose Solution
  Interventions: Device: O2Optix contact lens; Device: ReNu MultiPlus Multi-Purpose Solution
- Proclear CL and ReNu MPS with SICS (Other): Proclear contact lens and ReNu MultiPlus Multi-Purpose Solution
  Interventions: Device: Proclear contact lens; Device: ReNu MultiPlus Multi-Purpose Solution
- 02Optix CL and Clear Care LCS with SICS (Other): O2Optix contact lens and Clear Care lens care solution subject
  Interventions: Device: O2Optix contact lens; Device: Clear Care Cleaning and Disinfecting Solution
- Proclear CL and Clear Care LCS with SICS (Other): Proclear contact lens and Clear Care lens care solution
  Interventions: Device: Proclear contact lens; Device: Clear Care Cleaning and Disinfecting Solution
- 02Optix CL and ReNu MPS without SICS (Other): O2Optix contact lens and ReNu MultiPlus Multi-Purpose Solution
  Interventions: Device: O2Optix contact lens; Device: ReNu MultiPlus Multi-Purpose Solution
- Proclear CL and ReNu MPS without SICS (Other): Proclear contact lens and ReNu MultiPlus Multi-Purpose Solution
  Interventions: Device: Proclear contact lens; Device: ReNu MultiPlus Multi-Purpose Solution
- 02Optix CL and Clear Care LCS without SICS (Other): O2Optix contact lens and Clear Care lens care solution
  Interventions: Device: O2Optix contact lens; Device: Clear Care Cleaning and Disinfecting Solution
- Proclear CL and Clear Care LCS without SICS (Other): Proclear contact lens and Clear Care lens care solution
  Interventions: Device: Proclear contact lens; Device: Clear Care Cleaning and Disinfecting Solution

INTERVENTIONS:
Device: O2Optix contact lens — control contact lens to be worn daily for approximately 7 months for entire length of study.
  Arms: 02Optix CL and Clear Care LCS with SICS; 02Optix CL and Clear Care LCS without SICS; 02Optix CL and ReNu MPS with SICS; 02Optix CL and ReNu MPS without SICS
Device: Proclear contact lens — control contact lens to be worn for entire length of study.
  Arms: Proclear CL and Clear Care LCS with SICS; Proclear CL and Clear Care LCS without SICS; Proclear CL and ReNu MPS with SICS; Proclear CL and ReNu MPS without SICS
Device: ReNu MultiPlus Multi-Purpose Solution — lens solution for overnight lens disinfection
  Arms: 02Optix CL and ReNu MPS with SICS; 02Optix CL and ReNu MPS without SICS; Proclear CL and ReNu MPS with SICS; Proclear CL and ReNu MPS without SICS
Device: Clear Care Cleaning and Disinfecting Solution — lens solution for overnight lens disinfection
  Arms: 02Optix CL and Clear Care LCS with SICS; 02Optix CL and Clear Care LCS without SICS; Proclear CL and Clear Care LCS with SICS; Proclear CL and Clear Care LCS without SICS

SUMMARY:
The purpose of this study is to compare two marketed contact lens care solutions in regards to comfort and ocular health.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old.
* Signed Informed Consent and Investigator to record this on Case Report Form (CRF) in appropriate space.
* Require a visual correction in both eyes (monovision allowed but not monofit).
* Have a contact lens spherical distance requirement between +6.00D and -9.00D in both eyes.
* Astigmatism of 1.00D or less in the better eye and 1.50D or less in the other eye.
* Be correctable to a visual acuity of 20/30 (6/9) or better in each eye.
* Have normal eyes with no evidence of abnormality or disease.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Clinically significant corneal edema, corneal vascularisation, tarsal abnormalities, bulbar injection or any other abnormality of the cornea that would contraindicate contact lens wear.
* Worn lenses on an extended wear basis in the last 3 months.
* Diabetic.
* Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* Polymethyl methacrylate (PMMA) or rigid gas-permeable (RGP) lens wear in the previous 8 weeks.
* Has had refractive surgery. Has had eye injury/surgery within 8 weeks immediately prior to enrolment for this study.
* Abnormal lacrimal secretions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - North Little Rock, Arkansas
  - Campbell, California
  - Cupertino, California
  - Laguna Niguel, California
  - Mission Viejo, California
  - San Clemente, California
  - Colorado Springs, Colorado
  - Bloomington, Illinois
  - Neodesha, Kansas
  - Raytown, Missouri
  - Warrensburg, Missouri
  - Florence, New Jersey
  - Chagrin Falls, Ohio
  - Warren, Ohio
  - Kittanning, Pennsylvania
  - Moon Township, Pennsylvania
  - Nanticoke, Pennsylvania
  - State College, Pennsylvania
  - Warwick, Rhode Island
  - Chamberlain, South Dakota
  - Bartlett, Tennessee
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Midlothian, Virginia
  - Virginia Beach, Virginia
- Aston Triangle, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in both the US and UK and were screened, randomized, and assigned to a study arm.
Pre-assignment Details: A total of 473 subjects were attempted to be enrolled. There were 27 disqualified, 2 due to incorrect care system, 1 due to non-compliance, and 24 due to non-compliance from investigator, leaving 446 subjects recruited to participate.Of those remaining, 21 failed to meet inclusion or were excluded for a total of 425 subjects who started the study.
Groups:
- 02Optix CL and ReNu MPS: O2Optix contact lens and ReNu MultiPlus Multi-Purpose Solution
- Proclear CL and ReNu MPS: Proclear contact lens and ReNu MultiPlus Multi-Purpose Solution
- 02Optix CL and Clear Care LCS: O2Optix contact lens and Clear Care lens care solution
- Proclear CL and Clear Care LCS: Proclear contact lens and Clear Care lens care solution
Period: Phase 1 (Baseline to 4 Weeks)
Arm/Group | 02Optix CL and ReNu MPS | Proclear CL and ReNu MPS | 02Optix CL and Clear Care LCS | Proclear CL and Clear Care LCS
Started | 121 | 103 | 115 | 107
Completed | 117 | 100 | 103 | 105
Not Completed | 4 | 3 | 12 | 2
Not completed — Pregnancy | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — poor vision | 0 | 0 | 3 | 0
Not completed — poor comfort | 1 | 1 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Phase 2 (4 Weeks to 24 Weeks)
Arm/Group | 02Optix CL and ReNu MPS | Proclear CL and ReNu MPS | 02Optix CL and Clear Care LCS | Proclear CL and Clear Care LCS
Started | 117 | 100 | 103 | 105
Completed | 101 | 91 | 94 | 100
Not Completed | 16 | 9 | 9 | 5
Not completed — Adverse Event | 2 | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Poor vision | 1 | 1 | 1 | 0
Not completed — Poor comfort | 1 | 4 | 0 | 3
Not completed — Randomization strata filled | 9 | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clear Care LCS: Subjects assigned to Clear Care lens care solution
- ReNU MPS: Subjects assigned to ReNU multi purpose solution
- Total: Total of all reporting groups
Arm/Group | Clear Care LCS | ReNU MPS | Total
Number analyzed (Participants) | 208 | 217 | 425
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (11.8) | 33.4 (11.3) | 33.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 150 | 304
  Male | 54 | 67 | 121
Region of Enrollment [Number; unit: participants]
  United States | 189 | 198 | 387
  United Kingdom | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Wear Time
Description: Average hours per day that contact lens were worn.
Time Frame: 24 weeks
Population: Subjects included in analysis were those who completed the study and had complete data available for statistical analysis.
Measure: Least Squares Mean (Standard Error); unit: Hours
Groups:
- Clear Care Lens Cleaning Solution (LCS): All subjects assigned to Clear Care LCS
- ReNU Multi Purpose Solution (MPS): All subjects assigned to ReNU MPS
Arm/Group | Clear Care Lens Cleaning Solution (LCS) | ReNU Multi Purpose Solution (MPS)
Number analyzed (Participants) | 194 | 192
Hours | 13.57 (0.23) | 13.30 (0.23)

2. Primary Outcome: Average Daily Comfortable Wear Time
Description: Average hours per day that contact lens were worn comfortably.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Hours | 11.96 (0.29) | 11.39 (0.29)

3. Primary Outcome: Lens Comfort
Description: Lens comfort at time of month 6 visit, using a scale of 0 to 10, where 10=excellent.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
units on a scale | 8.63 (0.13) | 8.25 (0.13)

4. Primary Outcome: Frequency of Eye Discomfort
Description: Subjective measure of typical daily eye discomfort reported at month 6 visit using a scale of 0 to 3. 0=Never, 1=Infrequently, 2=Frequently, 3=Constantly.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
units on a scale | 0.36 (0.05) | 0.46 (0.05)

5. Primary Outcome: Frequency of Daily Lens Dryness
Description: Subjective measure of typical daily contact lens dryness reported at month 6 visit using a scale of 0 to 3. 0=Never, 1=Infrequently, 2=Frequently, 3=Constantly.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
units on a scale | 0.66 (0.05) | 0.68 (0.05)

6. Primary Outcome: Frequency of Eye Burning/Stinging
Description: Subjective measure of typical daily eye burning and stinging reported at month 6 visit using a scale of 0 to 3. 0=Never, 1=Infrequently, 2=Frequently, 3=Constantly.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
units on a scale | 0.31 (0.04) | 0.31 (0.04)

7. Primary Outcome: Frequency of Itching
Description: as for outcome 6
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Clear Care LCS: O2Optix contact lens and ReNu MultiPlus Multi-Purpose Solution
- ReNU MPS: Proclear contact lens and ReNu MultiPlus Multi-Purpose Solution
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
units on a scale | 0.21 (0.03) | 0.21 (0.03)

8. Primary Outcome: Frequency of Tearing
Description: Subjective measure of typical daily tearing related to lens wear reported at month 6 visit using a scale of 0 to 3. 0=Never, 1=Infrequently, 2=Frequently, 3=Constantly.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
units on a scale | 0.16 (0.03) | 0.15 (0.03)

9. Primary Outcome: Average Corneal Fluorescein Type Staining
Description: staining measured over five sectors of the cornea and classified as a type of staining on a scale of 0 to 4. 0=None, 1=Micropunctate, 2=Macropunctate, 3=Coalesced Macropunctate, 4=Patch.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (Eyes) | 388 | 384
units on a scale | 0.16 (0.02) | 0.36 (0.02)

10. Primary Outcome: Average Corneal Fluorescein Staining Area
Description: corneal staining measured over 5 areas, averaged, and graded as a single score average on a scale of 0 to 10, 0=0%, 1=10%, 2=20%, 3=30%, 4=40%, 5=50%, 6=60%, 7=70%, 8=80%, 9=90%, 10=100%.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (Eyes) | 388 | 384
units on a scale | 0.27 (0.09) | 0.99 (0.09)

11. Primary Outcome: Limbal Redness
Description: Redness at the transition zone between the white of the eye and the clear window of the eye, the cornea, on a scale of 0 to 4. 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (eyes) | 388 | 384
units on a scale | 0.44 (0.03) | 0.49 (0.03)

12. Primary Outcome: Bulbar Redness
Description: Redness of the blood vessels in the tissues overlaying the white of the eye, on a scale of 0 to 4. 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (eyes) | 388 | 387
units on a scale | 0.50 (0.03) | 0.56 (0.03)

13. Primary Outcome: Lower Tarsal Redness
Description: Redness of the blood vessels in the inner lining of the lower eyelid, on a scale of 0 to 4. 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (eyes) | 388 | 384
units on a scale | 0.51 (0.03) | 0.57 (0.03)

14. Primary Outcome: Upper Tarsal Redness
Description: Redness of the blood vessels in the inner lining of the upper eyelid, on a scale of 0 to 4. 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (eyes) | 388 | 384
units on a scale | 0.48 (0.03) | 0.55 (0.03)

15. Primary Outcome: Tarsal Roughness
Description: The roughness of the inner lining of the eyelids, measured on a 0 to 7 scale. 0=Smooth, 1=Slightly uneven, 2=Uneven surface, 3=Uneven surface with loss of transparency & superficial vessels, 4=Small papillae, poor transparency, 5=Papillae greater than 0.5mm in size, no transparency, 6=Papillae greater than 0.5mm in size, vessels inside papillae, 7=Large papillae
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Clear Care LCS | ReNU MPS
Number analyzed (Participants) | 194 | 192
Number analyzed (eyes) | 388 | 384
units on a scale | 0.75 (0.05) | 0.87 (0.05)

16. Secondary Outcome: Intensity of Physiological Outcomes
Description: Mean of physiological outcomes for those subjects who are identified as susceptible versus non-susceptible to "Solution Induced Corneal Staining (SICS)". These measures are related to intensity of outcomes, i.e. discomfort, burning, dryness, etc. with lower scores being better on a scale of 1-5.
Time Frame: 24 weeks
Population: All subjects, enrolled, randomized, and completed the study. Subjects where identified as 'stainers' or 'non-stainers' and outcomes were reported per this stratification.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- Clear Care LCS (Stainers); Clear Care LCS (Non-Stainers): Clear Care LCS users: Any subject that presented with diffuse punctate staining in three or more peripheral sectors in each eye was classified as a 'stainer' during slit-lamp examination, those who did not were termed 'non-stainers'.
- ReNU MPS (Stainers); ReNU MPS (Non-Stainers): ReNU users: Any subject that presented with diffuse punctate staining in three or more peripheral sectors in each eye was classified as a 'stainer' during slit-lamp examination, those who did not were termed 'non-stainers'.
Arm/Group | Clear Care LCS (Stainers) | Clear Care LCS (Non-Stainers) | ReNU MPS (Stainers) | ReNU MPS (Non-Stainers)
Number analyzed (Participants) | 78 | 116 | 69 | 123
units on a scale
  Intensity of Discomfort/Pain | 2.00 (1.22) | 2.41 (1.14) | 2.48 (1.09) | 2.24 (1.17)
  Intensity of Burning/Stinging | 2.24 (1.30) | 2.10 (1.16) | 2.35 (1.09) | 1.76 (1.00)
  Intensity of Dryness | 2.20 (0.95) | 2.69 (1.18) | 2.40 (1.06) | 2.25 (1.14)
  Intensity of Itching | 1.94 (0.93) | 1.70 (1.10) | 2.24 (1.23) | 1.67 (0.84)
  Intensity of Tearing | 2.00 (1.13) | 1.61 (0.78) | 2.38 (1.04) | 1.73 (0.79)

17. Secondary Outcome: Wearing Time and Comfortable Wearing Time
Description: Mean of physiological outcomes for those subjects who are identified as susceptible versus non-susceptible for "Solution Induced Corneal Staining (SICS)". Average wearing time and average comfortable wearing time.
Time Frame: 24 weeks
Population: as for outcome 16
Measure: Least Squares Mean (Standard Deviation); unit: hours
Arm/Group | Clear Care LCS (Stainers) | Clear Care LCS (Non-Stainers) | ReNU MPS (Stainers) | ReNU MPS (Non-Stainers)
Number analyzed (Participants) | 78 | 116 | 69 | 123
hours
  Average Wearing Time | 14.06 (2.24) | 13.63 (2.55) | 13.49 (2.67) | 13.33 (2.28)
  Average Comfortable Wearing Time | 12.42 (3.17) | 11.93 (3.47) | 11.35 (3.35) | 11.75 (3.67)

18. Secondary Outcome: Physiological Responses
Description: Mean of physiological outcomes for those subjects who are identified as susceptible versus non-susceptible for "Solution Induced Corneal Staining (SICS)". Physiological findings are done through a slit lamp examination and are known as biomicroscopy measurements. Measures are given in terms of average score with a minimum of zero and a worse grade the higher the value with a range of 0 to 4, (tarsal roughness is 0-7 scale).
Time Frame: 24 weeks
Population: All subjects, enrolled, randomized, and completed the study. Subjects where identified as 'stainers' or 'non-stainers' and outcomes were reported by this stratification.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clear Care LCS (Stainers) | Clear Care LCS (Non-Stainers) | ReNU MPS (Stainers) | ReNU MPS (Non-Stainers)
Number analyzed (Participants) | 78 | 116 | 69 | 123
units on a scale
  Corneal Staining | 0.20 (0.25) | 0.11 (0.19) | 0.52 (0.56) | 0.32 (0.38)
  Limbal Hyperemia | 0.52 (0.66) | 0.39 (0.50) | 0.46 (0.58) | 0.43 (0.51)
  Bulbar Hyperemia | 0.51 (0.59) | 0.48 (0.54) | 0.53 (0.62) | 0.52 (0.59)
  Lower Tarsal Hyperemia | 0.50 (0.63) | 0.48 (0.54) | 0.55 (0.68) | 0.59 (0.61)
  Upper Tarsal Hyperemia | 0.51 (0.60) | 0.46 (0.54) | 0.51 (0.60) | 0.59 (0.61)
  Tarsal Roughness | 0.97 (0.74) | 0.69 (0.75) | 0.90 (0.77) | 0.84 (0.89)

ADVERSE EVENTS:
Groups:
- Proclear CL and ReNu MPS: Proclear contact lens and ReNu MultiPlus Multi-Purpose
Arm/Group | 02Optix CL and ReNu MPS | Proclear CL and ReNu MPS | 02Optix CL and Clear Care LCS | Proclear CL and Clear Care LCS
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/103 | 0/115 | 1/107
Other Adverse Events (participants affected / at risk) | 0/121 | 0/103 | 0/115 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 02Optix CL and ReNu MPS (N=121) | Proclear CL and ReNu MPS (N=103) | 02Optix CL and Clear Care LCS (N=115) | Proclear CL and Clear Care LCS (N=107)
Viral Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written consent of the sponsor is required for publication.